CLINICAL TRIAL: NCT04393688
Title: A Prospective, Multicenter, Randomized, Controlled Study to Evaluate the Safety and Efficacy of a Tri-wire Balloon Dilatation Catheter for the Treatment of Dysfunctional AV Fistula
Brief Title: Study Evaluating the Safety and Efficacy of Tri-wire Balloon for Treatment of Dysfunctional AV Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BrosMed Medical Co., Ltd (Industry)
Collaborators: CCRF Inc., Beijing, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM-821
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Tri-wire Peripheral Balloon Dilatation Catheter (Experimental): Percutaneous transluminal angiography (PTA) will be performed using the Tri-wire Peripheral Balloon Dilatation Catheter. Interventions: Combination Product: Tri-wire Peripheral Balloon Dilatation Catheter; Procedure: Percutaneous Transluminal Angiography.
  Interventions: Combination Product: Combination Product: Tri-wire Peripheral Balloon Dilatation Catheter
- Active Comparator: OHICHO Ⅱ PTA Balloon Catheter. (Active Comparator): Percutaneous transluminal angiography (PTA) will be performed using OHICHO Ⅱ PTA Balloon Catheter, a commercially available high-pressure PTA balloon. Multiple balloons, inflations and/or prolonged inflation may be used. Interventions: Device: OHICHO Ⅱ PTA Balloon Catheter. Procedure: Percutaneous Transluminal Angiography.
  Interventions: Combination Product: Combination Product: Tri-wire Peripheral Balloon Dilatation Catheter

INTERVENTIONS:
Combination Product: Combination Product: Tri-wire Peripheral Balloon Dilatation Catheter — Procedure:
  Percutaneous Transluminal Angiography, Percutaneous transluminal angioplasty (PTA) is a procedure that can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored.
  Other Names: Device: OHICHO Ⅱ PTA Balloon Catheter

SUMMARY:
This prospective, multicenter, randomized, controlled study is designed to evaluate the safety and effectiveness of the Tri-wire Peripheral Balloon Dilatation Catheter compared to a standard PTA Catheter in treating subjects presenting with clinical and hemodynamic abnormalities in native arteriovenous (AV) fistulae located in the upper extremity.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years;
2. Able to understand the purpose of the study, willing to participate and sign the informed consent, able and willing to accept the follow-up;
3. Indications of percutaneous transluminal angioplasty for target lesion: target lesion shows >50% narrowing relative to adjacent normal vein diameter by angiography or ultrasound with one of the indicators listed in KDOQI vascular access guideline 2019 update Table 13.2.
4. Reference vessel diameter of target lesion from 3.0 mm to 8.0 mm.
5. Target lesion located from proximal to the anastomosis to the reflux vein at the distal end of the subclavian vein.
6. De novo or restenosis lesion.
7. Single or tandem lesion, length of which ≤ 60mm.

Exclusion Criteria:

1. Women who are pregnant, nursing, or planning to become pregnant during the study.
2. Patients who have accepted major surgeries within 30 days prior to the enrollment. (such as thoracic surgery, cranial surgery).
3. Patients who plan to accept major surgeries within 30 days after the enrollment. (such as thoracic surgery, cranial surgery).
4. Occlusion lesion or thrombosis.
5. Infected fistula or severe systemic infection.
6. Patients who suffer from central venous diseases.
7. Patients known to be allergic or contraindicated to contrast agents.
8. Patients who have participated in another clinical trial within 3 months prior to the study, or previous enrollment in this study.
9. Subject has another medical condition, which, in the opinion of the Investigator, may cause him/her to be noncompliant with the protocol or confound the data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Right after operation
  The target lesion residual stenosis<30%

SECONDARY OUTCOMES:
Device Success | Right after operation
  During the operation, Balloon dilatation catheters can be delivered to the target lesion, inflated≤RBP without rupture and withdrawed successfully
Procedural Success | 12-48 hours
  Base on the technical success, without MAE including death, thrombosis, allergic reactions, pulmonary diseases (pulmonary edema)
Dilating Pressure | During the operation
  The minimum pressure with which the balloon can be completely inflated without waist during the operation
Pain Score | Right after operation
  The pain during dilating procedure, measured by NRS (increase from 0 to 10)
Target Lesion Primary Patency (TLPP) | 1 month
  Defined as the interval following index procedure intervention until clinically driven reintervention of the target lesion or access thrombosis. TLPP ends with a clinically driven re-intervention of the target lesion or access thrombosis.
Target lesion restenosis | 1 month
  Target lesion diameter restenosis rate（measured by DUS）=100%*(1-(MLD/RVD)) (MLD includes 5mm range of proximal and distal of targer lesions
Fistula Blood Flow | 1 month
  Measured Brachial artery blood flow of arteriovenous fistula flow assessed by DUS.
Adverse Events | 1 month
  Number of device and procedure related adverse events (CEC Adjudicated)

CONTACTS AND LOCATIONS:
Overall Officials: Qizhuang Jin, Principal Investigator — Peking University First Hospital
Locations (7):
- China (7):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhengjiang

IPD SHARING:
Plan to Share IPD: No